CLINICAL TRIAL: NCT05867485
Title: The Effect of Special Discharge Training Prepared for Geriatric Patients in the COVID-19 Service on Daily Life Activities and Quality of Life
Brief Title: The Effect of Special Discharge Training in the COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kilis 7 Aralik University (Other)
Responsible Party: Principal Investigator, İslam Elagöz, Research Assıstant, Kilis 7 Aralik University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: AralikKilisU1
Record Dates: First submitted 2023-05-17; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Pneumonia
Keywords: COVID-19; Special Discharge Training; Geriatric; Daily Life Activities; Quality of Life
MeSH Terms: conditions — COVID-19 | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group: (No Intervention): Initially, the Patient Diagnostic Information Form was completed. Patients were informed about the discharge process according to the regular ward procedure and were informed about their participation in the study after discharge.
  One month later, patients were contacted by phone, and the Daily Life Activities Scale (DLAS) and Quality of Life Scale (SF-12) forms were completed during 10-15 minute conversations.
- Study Group: (Experimental): After obtaining informed consent from the patients, they were enrolled in the study.
  The COVID-19 Discharge Education Brochure, prepared by the researchers, was provided to the patients face-to-face within 10-15 minutes.
  One month after the discharge education, patients were contacted by phone, and the Daily Life Activities Scale (DLAS) and Quality of Life Scale (SF-12) forms were completed.
  Interventions: Other: COVID-19 Discharge Education

INTERVENTIONS:
Other: COVID-19 Discharge Education — A discharge education brochure has been developed based on information from the literature to complement the verbal information provided to patients. The content of the education brochure includes the following:
  1. Information about the spread of the virus and precautions to be taken.
  2. Guidelines for cleanliness and disinfection of the environment.
  3. Precautions regarding personal and wearable items.
  4. Information about food and beverages.
  5. Guidelines for personal hygiene practices.
  6. Information about quarantine and isolation.
  7. Guidelines for maintaining health and care (e.g., respiratory hygiene, cough etiquette, movement, range of motion exercises) (CDC, 2019; Ministry of Health of Turkey, 2020; CDC 2019 A-B-C-D).
  Other Names: education
  Arms: Study Group:

SUMMARY:
This study aimed to evaluate the impact of specialized discharge education on the daily life activities and quality of life of geriatric patients hospitalized in COVID-19 wards. The motivation behind this study stems from the vulnerability of elderly patients during the COVID-19 pandemic and the necessity of tailored education to support their daily life activities and enhance their quality of life after discharge. The primary objective of this article is to determine the specific type of specialized discharge education that geriatric patients in COVID-19 wards require to improve their ability to sustain daily life activities and enhance their quality of life.

The central idea of this study is that providing specialized discharge education to geriatric patients in COVID-19 wards can result in improvements in their daily life activities and quality of life. The main findings of the study demonstrate a significant enhancement in daily life activities and quality of life among patients who received specialized discharge education. These individuals exhibited increased independence in mobility, improved performance in daily life activities, and reported an overall improvement in their quality of life.

These findings underscore the significance of specialized discharge education for geriatric patients hospitalized in COVID-19 wards and highlight its positive impact on their health outcomes and quality of life.

DETAILED DESCRIPTION:
Purpose: This research aimed to determine the impact of specialized discharge training on the daily living activities and quality of life of geriatric patients admitted to the COVID-19 ward.

Materials and Methods: A quasi-experimental study was conducted on geriatric patients admitted to a training and research hospital's COVID-19 ward between April 1 and July 1, 2022. A control group of 40 individuals and a study group of 40 individuals, both meeting the inclusion criteria, were established. Research data were collected using the Descriptive Features Form, Katz Index of Independence in Activities of Daily Living, and SF-12 Quality of Life Scale.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the study were as follows; Willingness to participate in the research, Age 65 and over, Hospitalized geriatric patients in the pandemic service, Openness to communication and cooperation, Sound mental health, Absence of sensory impairments such as vision, hearing, and speech.

Exclusion Criteria:

* patients who do not meet the inclusion criteria

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Katz Daily Life Activities Scale (GYA): | 0 day
  The Katz Daily Life Activities Scale (GYA) was developed by Katz and colleagues in 1963 to assess activities essential for daily life. The scale measures the scores of key elements related to daily life activities, such as bathing, dressing, toileting, mobility, continence, and feeding. The GYA index categorizes scores as dependent (0-6 points), partially dependent (7-12 points), and independent (13-18 points). The scale has been translated into Turkish and validated by Yardımcı E., with a Cronbach's alpha coefficient of 0.73. Response options in the Katz GYA scale include "independent," "partially dependent," and "dependent."
Quality of Life Scale (SF-12): | 0 day
  The SF-12 Quality of Life Scale is a widely used instrument that assesses the quality of life over the past four weeks, encompassing various age and disease groups. The Turkish version of the scale, including its reliability and validity study, was conducted by Soylu and Kütük (2022). The SF-12 consists of 12 questions selected from the SF-36 Quality of Life Scale. It comprises eight sub-dimensions and 12 items, including physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The SF-12 yields two summary scores: the Physical Component Summary Score (PCSS) and the Mental Component Summary Score (MCSS). The scale demonstrates a Cronbach's alpha coefficient of 0.72.
Katz Daily Life Activities Scale (GYA): | 1 month
  The Katz Daily Life Activities Scale (GYA) was developed by Katz and colleagues in 1963 to assess activities essential for daily life. The scale measures the scores of key elements related to daily life activities, such as bathing, dressing, toileting, mobility, continence, and feeding. The GYA index categorizes scores as dependent (0-6 points), partially dependent (7-12 points), and independent (13-18 points). The scale has been translated into Turkish and validated by Yardımcı E., with a Cronbach's alpha coefficient of 0.73. Response options in the Katz GYA scale include "independent," "partially dependent," and "dependent."
Quality of Life Scale (SF-12): | 1 month
  The SF-12 Quality of Life Scale is a widely used instrument that assesses the quality of life over the past four weeks, encompassing various age and disease groups. The Turkish version of the scale, including its reliability and validity study, was conducted by Soylu and Kütük (2022). The SF-12 consists of 12 questions selected from the SF-36 Quality of Life Scale. It comprises eight sub-dimensions and 12 items, including physical functioning, physical role, bodily pain, general health, vitality, social functioning, emotional role, and mental health. The SF-12 yields two summary scores: the Physical Component Summary Score (PCSS) and the Mental Component Summary Score (MCSS). The scale demonstrates a Cronbach's alpha coefficient of 0.72.

CONTACTS AND LOCATIONS:
Overall Officials: islam ELAGÖZ, PhD-c, Principal Investigator — Kilis yesi Aralık Universty
Locations (1):
- Islam, Kilis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No